CLINICAL TRIAL: NCT00015002
Title: A Randomized Placebo-Controlled Trial of Antenatal Corticosteroid Regimens
Brief Title: Repeat Antenatal Steroids Trial
Acronym: BEARS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Concerns regarding neonatal data
Sponsor: The George Washington University Biostatistics Center (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Treatment
Other Study IDs: NICHD-0801; HD21410; HD27869; HD27917; HD27860; HD27915; HD34116; HD34208; HD34136; HD40500; HD40485; HD40544; HD40545; HD40560; HD40512; HD36801
Record Dates: First submitted 2001-04-17; First posted 2001-04-18 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Complications, Pregnancy
Keywords: Antenatal corticosteroids; Preterm delivery
MeSH Terms: conditions — Pregnancy Complications; Premature Birth | interventions — Betamethasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Betamethasone — coded study medication is 12 mg of betamethasone (or placebo) given as 2 ml intramuscular injection in 2 doses, 24 hours apart (the "Course"). Patients administered weekly courses for 4 weeks, until 33 weeks 6 days gestation or delivery, whichever occurs first.

SUMMARY:
A course of steroids given to a mother who is in labor with a premature fetus will reduce the risk of the premature infant dying or having serious complications. This trial will test whether more than one course of antenatal steroids is more beneficial or risky to the infant than a single course.

DETAILED DESCRIPTION:
After the NICHD Consensus Development Conference in 1994, the antenatal administration of antenatal corticosteroids (betamethasone or dexamethasone) for prevention of death and the serious morbidities associated with preterm birth has become an accepted standard in American obstetric practice. Studies have shown that maximum beneficial effect occurs when the fetus is delivered within 7 days of antenatal steroid administration. The efficacy and safety of a single course of corticosteroids has been substantiated but it is unknown whether repetitive dosing has similar efficacy or what the maternal, fetal and neonatal risks are. Repeat courses of steroids are often administered. Two popular regimens exist for the patient who remains undelivered more than one week after initial therapy but who remains at risk for preterm birth. In one, steroids are repeated weekly until 34 weeks gestation, while in the other, steroids are only given once.

This multicenter trial is testing the safety and efficacy of weekly administration of antenatal steroids. Twenty four hundred women < 32.0 weeks gestation who are at risk for spontaneous preterm delivery and remain pregnant at least seven days after an initial course of corticosteroids are being randomized to either weekly courses of masked study drug (betamethasone or placebo) for 4 weeks or delivery, whichever comes first. Patients are asked about side effects at the weekly visits and samples of maternal blood at randomization and delivery are collected. Cord blood and placentas are also collected. Cranial ultrasounds are done on all neonates. On a subgroup of patients, an adrenocorticotrophic hormone (ACTH) stimulation test is being performed and an auditory brainstem response (ABR) performed. All infants attend a follow-up visit at 18 to 22 months corrected age where certified examiners, masked to study group assignment, collect physical and neurological data. The Bayley Scales of Infant Development will also be administered. A subgroup of infants will be seen at 36 months to administer the Intelligence scale from the McCarthy Scales of Children's Abilities.

ELIGIBILITY:
Inclusion criteria:

* Pregnant
* Gestational age > 23.0 wks and < 31.6 wks
* Singleton or twin pregnancy
* Intact membranes
* At-risk for spontaneous preterm delivery
* Received full course of corticosteroids within the previous 7 days

Exclusion criteria:

* Diagnosis of fetal lung maturity
* Chorioamnionitis
* Non-reassuring fetal testing
* Known major fetal anomaly
* Corticosteroid therapy, other than qualifying course
* Insulin dependent diabetes
* Active preterm labor at the time of randomization
* Delivery intended outside center
* Participation in any intervention study which influences neonatal morbidity or mortality
* Previous participation in this trial

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 486 (Actual)
Dates: Start 2000-03; Primary Completion 2006-05 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
Composite outcome: including neonatal mortality/stillbirth, severe RDS, chronic lung disease, grade III/IV IVH, PVL

SECONDARY OUTCOMES:
Neonatal morbidity
Maternal morbidity
Neonatal Growth parameters
Infant neurological parameters

CONTACTS AND LOCATIONS:
Overall Officials: Ronald J Wapner, MD, Principal Investigator — MCP Hahnemann University Hospital
Locations (19):
- United States (19):
  - University of Alabama, Birmingham, Alabama
  - University of Miami, Miami, Florida
  - Northwestern University-Prentice Hospital, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Dept of OB/GYN, Hutzel Hospital, Detroit, Michigan
  - Columbia University, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Forsyth Memorial Hospital, Wake Forest University School of Medicine, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve-Metrohealth, Cleveland, Ohio
  - Dept of OB/GYN, Ohio State University, Columbus, Ohio
  - MCP Hahnamann, Philadelphia, Pennsylvania
  - Dept of OB/GYN, Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Brown University -Women and Infants Hospital, Providence, Rhode Island
  - University of Tennessee, Memphis, Tennessee
  - Dept of OB/GYN, Southwestern Medical Center, University of Texas, Dallas, Texas
  - University of Texas-Houston, Houston, Texas
  - University of Texas - San Antonio, San Antonio, Texas
  - University of Utah Medical Center, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
The data will be shared after completion and publication of the main analyses in accordance with NIH policy. The dataset can be obtained by emailing mfmudatasets@bsc.gwu.edu

REFERENCES:
- [Background] Liggins GC, Howie RN. A controlled trial of antepartum glucocorticoid treatment for prevention of the respiratory distress syndrome in premature infants. Pediatrics. 1972 Oct;50(4):515-25. No abstract available. PMID 4561295
- [Background] Crowley PA. Antenatal corticosteroid therapy: a meta-analysis of the randomized trials, 1972 to 1994. Am J Obstet Gynecol. 1995 Jul;173(1):322-35. doi: 10.1016/0002-9378(95)90222-8. No abstract available. PMID 7631713
- [Background] French NP, Hagan R, Evans SF, Godfrey M, Newnham JP. Repeated antenatal corticosteroids: size at birth and subsequent development. Am J Obstet Gynecol. 1999 Jan;180(1 Pt 1):114-21. doi: 10.1016/s0002-9378(99)70160-2. PMID 9914589
- [Background] Effect of corticosteroids for fetal maturation on perinatal outcomes. NIH Consensus Development Panel on the Effect of Corticosteroids for Fetal Maturation on Perinatal Outcomes. JAMA. 1995 Feb 1;273(5):413-8. doi: 10.1001/jama.1995.03520290065031. PMID 7823388
- [Background] Gamsu HR, Mullinger BM, Donnai P, Dash CH. Antenatal administration of betamethasone to prevent respiratory distress syndrome in preterm infants: report of a UK multicentre trial. Br J Obstet Gynaecol. 1989 Apr;96(4):401-10. doi: 10.1111/j.1471-0528.1989.tb02413.x. PMID 2665800
- [Background] Effect of antenatal dexamethasone administration on the prevention of respiratory distress syndrome. Am J Obstet Gynecol. 1981 Oct 1;141(3):276-87. PMID 7025638
- [Background] Wright LL. Evidence from multicenter networks on the current use and effectiveness of antenatal corticosteroids in very low birthweight infants. In: National Institute of Child Health and Development (US). Report on the Consensus Development Conference on the Effect of Corticosteroids for Fetal Maturation on Perinatal Outcomes; 1994 Feb 28-Mar 2; Bethesda, (MD): The Institute; 1994 Nov. P. 47-8. (NIH Publication; no. 95-3784).
- [Result] Wapner RJ, Sorokin Y, Thom EA, Johnson F, Dudley DJ, Spong CY, Peaceman AM, Leveno KJ, Harper M, Caritis SN, Miodovnik M, Mercer B, Thorp JM, Moawad A, O'Sullivan MJ, Ramin S, Carpenter MW, Rouse DJ, Sibai B, Gabbe SG; National Institute of Child Health and Human Development Maternal Fetal Medicine Units Network. Single versus weekly courses of antenatal corticosteroids: evaluation of safety and efficacy. Am J Obstet Gynecol. 2006 Sep;195(3):633-42. doi: 10.1016/j.ajog.2006.03.087. Epub 2006 Jul 17. PMID 16846587
- [Result] Carroll MA, Vidaeff AC, Mele L, Wapner RJ, Mercer B, Peaceman AM, Sorokin Y, Dudley DJ, Spong CY, Leveno KJ, Harper M, Caritis SN, Miodovnik M, Thorp JM, Moawad A, O'Sullivan MJ, Carpenter MW, Rouse DJ, Sibai B; National Institute of Child Health and Human Development (NICHD) Maternal Fetal Medicine Units Network (MFMU). Bone metabolism in pregnant women exposed to single compared with multiple courses of corticosteroids. Obstet Gynecol. 2008 Jun;111(6):1352-8. doi: 10.1097/AOG.0b013e318173573b. PMID 18515519
- [Result] Fonseca L, Ramin SM, Mele L, Wapner RJ, Johnson F, Peaceman AM, Sorokin Y, Dudley DJ, Spong CY, Leveno KJ, Caritis SN, Miodovnik M, Mercer B, Thorp JM, O'Sullivan MJ, Carpenter MW, Rouse DJ, Sibai B; Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) Maternal Fetal Medicine Units Network (MFMU). Bone metabolism in fetuses of pregnant women exposed to single and multiple courses of corticosteroids. Obstet Gynecol. 2009 Jul;114(1):38-44. doi: 10.1097/AOG.0b013e3181a82b85. PMID 19546756
- [Result] Sawady J, Mercer BM, Wapner RJ, Zhao Y, Sorokin Y, Johnson F, Dudley DJ, Spong CY, Peaceman AM, Leveno KJ, Harper M, Caritis SN, Miodovnik M, Thorp JM, Ramin S, Carpenter MW, Rouse DJ; National Institute of Child Health and Human Development Maternal Fetal Medicine Units Network. The National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network Beneficial Effects of Antenatal Repeated Steroids study: impact of repeated doses of antenatal corticosteroids on placental growth and histologic findings. Am J Obstet Gynecol. 2007 Sep;197(3):281.e1-8. doi: 10.1016/j.ajog.2007.06.041. PMID 17826421
- [Result] Wapner RJ, Sorokin Y, Mele L, Johnson F, Dudley DJ, Spong CY, Peaceman AM, Leveno KJ, Malone F, Caritis SN, Mercer B, Harper M, Rouse DJ, Thorp JM, Ramin S, Carpenter MW, Gabbe SG; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network. Long-term outcomes after repeat doses of antenatal corticosteroids. N Engl J Med. 2007 Sep 20;357(12):1190-8. doi: 10.1056/NEJMoa071453. PMID 17881751
- See also: Click here for more information on the NICHD MFMU Research Network. — http://www.bsc.gwu.edu/mfmu/